CLINICAL TRIAL: NCT00647140
Title: Clinical Evaluation of 18F-DOPA Positron Emission Tomography in Medullary Thyroid Cancer.
Acronym: DOPMET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insuffisent recruitment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Zakia.IDIR, Department Clinical Research of Developpemnt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P051081
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-05

CONDITIONS: Thyroid Neoplasm; Thyroid Carcinoma; Medullary Carcinoma
Keywords: Thyroid neoplasm; Thyroid carcinoma; Medullary carcinoma; Positron Emission Tomography (PET); 18F-L DOPA; Calcitonin; Carcinoembryonic Antibodies; Cervical ultrasonography; Cervical-chest-abdomen tomography; Cervical-chest-abdomen magnetic resonance imaging; Osseous radionuclide imaging; Post-PET surgery; Post-PET biopsy; Post-PET histology
MeSH Terms: conditions — Thyroid Neoplasms; Carcinoma, Medullary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 18F-L6DOPA PET
  Interventions: Other: 18F-L-DOPA PET

INTERVENTIONS:
Other: 18F-L-DOPA PET — PET performed 30 minutes after IV injection of 4 MBq/kg of 18F-DOPA
  Other Names: 18F-L-DOPA Positron Emission Tomography

SUMMARY:
Medullary thyroid carcinoma (MTC) is a rare tumor arising from C cells of the thyroid gland and belonging to the endocrine tumors. 18F-DOPA PET, based on tha capacity of endocrine tumor cells to take-up, decarboxylate and store amino-acids, such 3-4-dihydroxyphenylalanine(DOPA), is used for imaging endocrine tumors. The aim of the study was to evaluate the contribution of 18F-DOPA whole-body PET for the detection of recurrences in patients with proven recurrent MTC without evidence of recurrence or metastases on several imaging modalities.

DETAILED DESCRIPTION:
In patients MTC and persistently elevated calcitonin levels, the challenge is finding the site of residual disease. Since the only satisfying treatment is surgery, the early detection and precise location is important. Tumor localization techniques usually performed, including ultrasonography of the neck and liver, chest and abdomen, bone scintigraphy, isotopic scanning and even PET with FDG are poorly sensitive. The use of 18F-DOPA may be more sensitive and specific engineering for localization metastatic disease. The study include 100 patient with persistent MTC demonstrated by elevated tumor markers (calcitonin and CEA) and no evidence of recurrence on morphological imaging procedures. 18F-DOPA whole-body PET is performed 30 minutes after IV injection of 4 MBq/kg of 18F-DOPA, the patient fasted for 6 hours prior the start of the examination.

All 18F-DOPA PET are evaluated independently by two experienced nuclear medicine physicians and any tracer accumulation exceeding the normal uptake tissue is rated as pathologic finding. The sensibility and efficiency of 18F-DOPA PET will be analysed and Malignant tissue confirmed by histology after surgery or biopsy or by follow-up for one year.

ELIGIBILITY:
Inclusion criteria:

* Patients up to 18 years old with medullary thyroid cancer / carcinoma
* Patients with medullary thyroid cancer / carcinoma recurrence, which have a high calcitonin level / rate, more than 100pg/ml, associated - or not - to a high CEA (Carcinoembryonic Antibodies) level / rate, dated from less than 3 months
* Patients with a less than 3 months conventional imaging checkup (cervical ultrasonography, cervical-chest-abdomen tomography and / or magnetic resonance imaging, abdomen ultrasonography, osseous / bones radionuclide imaging), in which the tumor site not certainty located
* Informed Consent Form signed and dated by patients
* Patients which are "SECURITE SOCIALE" affiliated

Exclusion criteria:

* Pregnant or suckling women
* Women able to procreate, without efficient birth control
* Patients already included in another Nuclear Medicine or Imaging research protocol using ionizing radiations; the efficient dose accumulation will not exceed 20 mSv.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Any tracer accumulation exceeding the normal uptake tissue searched by two experienced nuclear medicine physicians and compared by malignant tissue confirmed by histology after biopsy, surgery or by follow-up for one year. | At the 18F-L-DOPA PET and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Badia-Ourkia HELAL, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris Hôpital Antoine Béclère
Locations (1):
- Hôpital Antoine Beclere, Clamart, France